CLINICAL TRIAL: NCT02919878
Title: Phase II Study of Neo-adjuvant Chemoradiotherapy Using Infusional Gemcitabine Followed by Surgery for Locally Advanced (T3 and T4 or Node Positive) Rectal Adenocarcinoma
Brief Title: Neo-adjuvant Chemoradiotherapy Using Infusional Gemcitabine Followed by Surgery for Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2141-124
Record Dates: First submitted 2015-03-24; First posted 2016-09-29 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Rectal Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pre-op Gemcitabine & XRT (Experimental): Pre-op chemo: Gemcitabine will be administered as continuous infusion IV over 24 hrs (100 mg/m2) weekly for 6 wks starting on day 1 of Radiotherapy (XRT).
  XRT/ Intensity modulated radiotherapy(IMRT): 1.8 Gy/fx, 5 fractions/wk will be delivered. Pelvis will receive 45 Gy/25 fractions/5 wks with a boost dose of 5.4 Gy for T3 and 9 Gy for T4 to a cone down volume. The total tumor dose= 50.4 -54 Gy.
  Post-op chemo: Standard 6 cycles of adjuvant Capecitabine (1250 mg/m2) PO twice per day on days 1-14 each cycle, (every 21 days) in patients who have a complete resection of rectal cancer and negative surgical margins.
  Interventions: Drug: Gemcitabine; Radiation: XRT; Drug: capecitabine

INTERVENTIONS:
Drug: Gemcitabine — Nucleoside analog- Chemotherapy
  Other Names: Gemzar
Radiation: XRT — pre-operative radiotherapy given concurrently with Gemcitabine chemotherapy
  Other Names: External beam radiotherapy (XRT)
Drug: capecitabine — Capecitabine is given post operatively as adjuvant chemotherapy for 6 cycles. Each cycle consist of 2500 mg/m2 per day given orally from D1-14
  Other Names: Xeloda

SUMMARY:
Phase II Study of Neo-adjuvant Chemoradiotherapy using infusional Gemcitabine followed by Surgery for Locally Advanced (T3 and T4 or Node positive) Rectal Adenocarcinoma.

DETAILED DESCRIPTION:
Results of neo-adjuvant chemo-radiation for advanced rectal cancer have plateaued with pathological complete response rates of 10-20% in spite of the addition of new cytotoxic agents and/ or molecular targeted therapies. The combination of 5-fluorouracil and radiation produces effective sensitization but further improvements require assessment of other sensitizers to increase the pathological complete response rates. Gemcitabine has been used in combination with radiation for several GI cancers but few studies have examined its role in rectal cancer. This study will examine a combination of Gemcitabine and radiation as neo-adjuvant therapy in advanced rectal cancer to increase the pathological complete response (pCR) rate from the investigators traditional 6% to > 40 %.

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma of the rectum without evidence of distant metastases
2. Patient must be 18 years of age or greater
3. Potentially resectable disease based upon surgeons evaluation
4. Clinical stages T3 or T4a, and/ or positive nodes based upon endorectal ultrasound and/ or MRI.
5. Absolute neutrophil count of > 1500 per microliter and platelet count > 100,000 per microliter; Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and alkaline phosphatase < 2.5 X upper limit of normal (ULN), bilirubin < = 1.5 ULN, calculated creatinine clearance > 50 ml/min using Cockcroft-Gault formula:

   Male: Creatinine Clearance = (140 - age) x weight/(72 X serum creatinine) Female: Creatinine Clearance = (140 - age) x weight/(72 X serum creatinine x 0.85)
6. Eastern cooperative oncology group (ECOG) performance status 0-2
7. No history of other malignancies within 5 years, except non-melanoma skin cancer, in situ carcinoma of the cervix, or ductal carcinoma in situ of the breast. Previous invasive cancer permitted if disease free at least 5 years.
8. Signed study-specific informed consent prior to enrolment

Exclusion Criteria:

1. Any evidence of distant metastasis
2. Synchronous primary colon carcinomas, except T1 lesions (full colonoscopy not required for enrollment)
3. Extension of malignant disease to the anal canal
4. Prior radiation therapy to the pelvis
5. Prior chemotherapy for malignancies
6. Pregnancy or lactation, (exclusion due to potential adverse effects of therapy). Women of childbearing potential with either a positive or no pregnancy test (serum or urine) at baseline. Women/men of childbearing potential not using a reliable and appropriate contraceptive method. (Postmenopausal women must have been amenorrheic for at least 12 months to be considered to be of non-childbearing potential.) Patients will agree to continue contraception for 30 days from the date of the last study drug administration.
7. Serious, uncontrolled, concurrent infection(s).
8. Participation in any investigational drug study within 4 weeks preceding the start of study treatment
9. Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
10. Evidence of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake
11. Other serious uncontrolled medical conditions that the investigator feels might compromise study participation.
12. Major surgery within 4 weeks of the study treatment
13. Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
14. Known, existing uncontrolled coagulopathy
15. No concurrent cimetidine allowed

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Estimate the rate of pathological complete response following neoadjuvant combined-modality therapy using weekly Gemcitabine and radiation therapy in rectal cancer. | "3 years"
  PCR will be assessed during the course of study

SECONDARY OUTCOMES:
Estimate the incidence of hematologic and non-hematologic grade 3-4 toxicity with the above regimen | "3 years"
  Toxicity will be evaluated for 3 years and beyond
Predictive value of positron Emission Tomography (PET) scan | within 2 month of finishing pre-operative chemoradiotherapy
  To assess the positive predictive value and negative predictive value of positive PET and negative PET for pathological complete response. In addition we will correlate the decrease of SUVmax by 50% with survival in patient treated with neo-adjuvant radiotherapy and Gemcitabine in for locally advanced rectal cancer
R0 resection rate | at the time of surgery ( 2.5 months) from completion of pre-operative chemoradiotherapy
  To assess the adequacy of R0 resection for tumors following down staging using the pre-operative concurrent chemoradiotherapy with Gemcitabine.

CONTACTS AND LOCATIONS:
Overall Officials: Shouki Bazarbashi, MD, Principal Investigator — KFSH&RC
Locations (1):
- Oncology Centre, King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bazarbashi S, Elshenawy MA, Badran A, Aljubran A, Alzahrani A, Almanea H, Alsuhaibani A, Alashwah A, Neimatallah M, Abduljabbar A, Ashari L, Alhomoud S, Ghebeh H, Elhassan T, Alsanea N, Mohiuddin M. Neoadjuvant concurrent chemoradiotherapy using infusional gemcitabine in locally advanced rectal cancer: A phase II trial. Cancer Med. 2022 May;11(10):2056-2066. doi: 10.1002/cam4.4590. Epub 2022 Feb 10. PMID 35146939